CLINICAL TRIAL: NCT00110565
Title: Pulsed Electromagnetic Field (PEMF) Efficacy in Reducing Rheumatoid Arthritis Symptoms
Brief Title: Effects of Pulsed Magnetic Pads on Rheumatoid Arthritis Symptoms in Postmenopausal Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R21AT001469-01A2 (NIH)
Record Dates: First submitted 2005-05-10; First posted 2005-05-11 (Estimated); Last update posted 2008-08-06 (Estimated); Status verified 2008-08

CONDITIONS: Rheumatoid Arthritis; Menopause
Keywords: Magnetics; Pulsed Magnetic Pad; Magnetic Field; Electromagnetic Field; Women; Pulsed Magnetic Field
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Pulsed magnetic field pad

SUMMARY:
The purpose of this study is to determine whether a pulsed magnetic field (PMF) pad will improve symptoms of rheumatoid arthritis (RA) in postmenopausal women.

Study hypothesis: A pulsed magnetic field pad will effectively reduce the symptoms of RA in postmenopausal women.

DETAILED DESCRIPTION:
RA is a condition characterized by pain, fatigue, sleep disturbances, and mood changes. These symptoms often persist despite the use of nonsteroidal anti-inflammatory drugs (NSAIDs) and disease modifying antirheumatic drugs (DMARDs). Many women for whom these drugs do not work turn to complementary and alternative therapies, including the use of magnetic devices. Although few studies have investigated the effects of low strength PMF pads in persons with RA, evidence suggests that PMF may help relieve pain, inflammation, and fatigue. This study will determine the effects of a PMF device on RA symptoms in postmenopausal women.

This study will last 12 weeks. Participants will be randomly assigned to one of three groups: active PMF pad treatment, sham PMF pad treatment, or standard of care, which may include drug therapy or physical therapy. Participants in the active and sham PMF pad groups will be treated with their assigned pad for approximately 8 minutes, twice a day for the duration of the study. Questionnaires and self-report scales will be used to assess pain, fatigue, sleep quality, mood, and inflammation episodes. Blood and urine collection will occur to assess levels of stress hormones and certain proteins.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of RA
* Postmenopausal, defined by no menstrual period in at least 2 years prior to study entry or a hysterectomy
* Average pain of 2 or greater on a 0 to 10 pain scale
* Sleep difficulty
* Stable medication use related to RA for at least 4 weeks prior to study entry

Exclusion Criteria:

* Diagnoses of lupus, sleep apnea, or restless leg syndrome
* High-dose prednisone (more than 10 mg/day) or equivalent
* Pacemakers or other implanted devices
* Epilepsy
* Currently undergoing treatment for cancer

Min Age: 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87
Dates: Start 2005-01; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Pain

SECONDARY OUTCOMES:
Fatigue
sleep disturbances
depression
perceived stress
stress hormones (norepinephrine and epinephrine)
cortisol
pro-inflammatory cytokines (IL-1, IL-6)
erythrocyte sedimentation rate (ESR)
C-reactive protein (CRP)
functional status
feasibility of study

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl M. Bourguignon, PhD, RN, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States